CLINICAL TRIAL: NCT03420365
Title: The Effect of a Single Bout of Aerobic Exercise Versus a Single Bout of Balance and Coordination Exercise on Cognitive Function in Elderly People
Brief Title: The Effect of a Single Bout of Balance and Coordination Exercise on Cognitive Function in Elderly People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: The Academic College at Wingate, Israel (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HYMC-0136-17
Record Dates: First submitted 2018-01-17; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Aging; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type of intervention (Experimental): A single bout of aerobic exercise, or a single bout of balance and coordination exercise, or reading a magazine
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — 30 minutes of either aerobic, or balance and coordination, or reading magazines
  Other Names: Balance and coordination exercise; Control

SUMMARY:
Individuals of advanced age are at higher risk of cognitive deterioration.A single bout of aerobic exercise was found to improve cognitive functions. The aim of this study is to explore the effect of a single bout of balance and coordination exercise versus aerobic exercise on cognitive functions among elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Able to undergo physical activity for 60 minutes
* Participates in a physical activity center at least twice a week

Exclusion Criteria:

* Scores beneath 24 on MMSE
* Unable to sign a consent form

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Cognitive function - Attention | Each cognitive test will be performed immediately following the intervention
  This cognitive domain will be based on scores of two tests: Go-NoGo test and the Stroop test, which will be performed by the use of NeuroTrax (NeuroTrax Corp., Israel) computerized battery that utilizes novel adaptations of traditional neuropsychological tests. In order to assess attention the mean reaction times (RTs) for the Go-NoGo test and the no-interference (meaning) phase of the Stroop test, and mean SD of RT for the Go-NoGo test will be calculated.
Cognitive function - Executive functions | Each cognitive test will be performed immediately following the intervention
  This cognitive domain will be based on scores of three tests: Go-NoGo test, Catch game and the Stroop test, which will be performed by the use of NeuroTrax (NeuroTrax Corp., Israel) computerized battery that utilizes novel adaptations of traditional neuropsychological tests. In order to assess executive function Performance indices for the Stroop test and the Go-NoGo test, and mean accuracy for the Catch Game will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- The Academic College at Wingate, Netanya, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol Statistical Analysis Plan